CLINICAL TRIAL: NCT03015168
Title: Prognostic Value of Neutrophil-to-lymphocyte Ratio (NLR) on Rectal Cancer Patients Who Received Capecitabine and Concurrent Intensity Modulated Radiotherapy (IMRT)
Brief Title: Prognostic Value of Neutrophil-to-lymphocyte Ratio (NLR) on Rectal Cancer Patients
Status: Completed | Type: Observational
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Radiation Oncology 201602
Record Dates: First submitted 2017-01-06; First posted 2017-01-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Rectal Cancer; Prognosis
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational Group: Patients with rectal cancer undergoing capecitabine and concurrent intensity modulated radiotherapy
  Interventions: Radiation: capecitabine and concurrent intensity modulated radiotherapy

INTERVENTIONS:
Radiation: capecitabine and concurrent intensity modulated radiotherapy — patients with rectal cancer undergoing capecitabine and concurrent intensity modulated radiotherapy

SUMMARY:
We explored the relationship between NLR and grade 3 or higher treatment related small bowel toxicity and treatment outcome of patients with rectal cancer undergoing capecitabine and concurrent intensity modulated radiotherapy (IMRT).

DETAILED DESCRIPTION:
Gender, age, stage of disease, and pathologic factors were retrospectively obtained from electronic patient records. Staging was determined according to the classification established by the American Joint Committee on Cancer (AJCC, 7th edition).Pelvic magnetic resonance imaging (MRI) were used for pretreatment staging. All patients enrolled in this study were treated with intensity modulated radiotherapy (IMRT) concurrent with capecitabine (1600 mg/m2/d, administered twice daily for two weeks) before or after curative resection. The mean radiation dose was 50 Gy with daily fraction of 2.0 Gy.

Acute treatment toxicity was scored according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE; version 3.0) and late toxicity was classified according to the Late Effects in Normal Tissue-Subjective, Objective, Management and Analytic (LENT-SOMA) system.

After the whole treatment procedure, all patients were subjected to a follow-up every three months for the first two years, every six months for the next three years, and every year thereafter. Physical examinations, routine blood test, serum carcinoembryonic antigen (CEA) and Cancer Antigen 19-9 (CA-199) level were checked at each follow up. Chest, abdominal CT scan and total colonoscopy were performed annually except the suspicion of tumor recurrence.

Overall survival (OS) time was defined from the date of completion of treatment to death from any cause and progression-free survival (PFS) time was defined as the time from the date of completion of therapy to the date of local recurrence or distant metastasis or death. Patient follow-up was lasted until death or the cutoff date of January 2017.Blood sampling reports from each enrolled patient were obtained within seven days before treatment. White blood cell count, neutrophil, lymphocyte and platelet counts were examined. The NLR was calculated as the absolute neutrophil count divided by the absolute lymphocyte count using baseline blood test results.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced rectal cancer who received neoadjuvant or adjuvant chemoradiotherapy at our hospital were enrolled in this study.

Exclusion Criteria:

* Patients with coexistent autoimmune diseases, infectious diseases, and lacking baseline blood test records were excluded from this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with rectal cancer undergoing capecitabine and concurrent intensity modulated radiotherapy
Sampling Method: Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2012-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
overall survival | 5years

SECONDARY OUTCOMES:
grade 3 or higher treatment related small bowel toxicity | 5years

CONTACTS AND LOCATIONS:
Overall Officials: Yan-Yang Wang, M.D., Principal Investigator — General Hospital of Ningxia Medical University
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: No